CLINICAL TRIAL: NCT05733234
Title: Lasers in Peri-implantitis Treatment YAG and Er: YAG Laser Approach, Investigation of Clinical and Bone Loss Biomarkers
Brief Title: Lasers in Peri-implantitis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Ioannis Fragkioudakis, Principal Investigator, Aristotle University Of Thessaloniki
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Frag2
Record Dates: First submitted 2023-01-19; First posted 2023-02-17 (Actual); Last update posted 2023-02-17 (Actual); Status verified 2023-02

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Test (Experimental): Laser-assisted surgical treatment of peri-implantitis
  Interventions: Device: Laser ,Fotona, Light Walker AT, Ljubljana, Slovenia
- Control (Active Comparator): Surgical treatment of peri-implantitis - No laser
  Interventions: Drug: Mechanical Treatment

INTERVENTIONS:
Device: Laser ,Fotona, Light Walker AT, Ljubljana, Slovenia — Laser is used adjunctively in the surgical treatment of peri-implantitis for decontamination of the implant surface
  Arms: Test
Drug: Mechanical Treatment — Dental instrument is used in combination with Chlorhexidine to decontaminate the implant surface
  Arms: Control

SUMMARY:
The current study aimed to investigate the effect of the combined Nd-Er: YAG laser on the surgical treatment of peri-implantitis by evaluating clinical markers and biomarkers of bone loss (RANKL/OPG). Twenty (20) patients having at least 1 implant diagnosed with peri-implantitis were randomly assigned to two groups for surgical treatment. In the test group (n=10), Er: YAG laser was used for granulation tissue removal and implant surface decontamination, while Nd: YAG laser was employed for deep tissue decontamination and biomodulation. In the control group (n=10), an access flap was applied, and mechanical instrumentation of the implant surface was performed by using titanium curettes. The following clinical parameters were evaluated at baseline and six months after treatment: Full-mouth Plaque Score (FMPS), Probing Pocket Depth (PPD), Probing Attachment Levels (PAL), recession (REC), and Bleeding on probing (BoP). Peri-implant crevicular fluid (PICF) was collected at baseline and six months for the evaluation of soluble RANKL and OPG utilizing enzyme-linked immunosorbent assay (ELISA).

DETAILED DESCRIPTION:
The study was designed as a prospective, randomized, controlled trial of a 6-month duration. Participants were recruited from the Department of Periodontology and Implant Biology of the Dental Faculty, School of Health Sciences, Aristotle University of Thessaloniki. Patients participating in this study should have at least one implant diagnosed with peri-implantitis according to the 2017 world Workshop on Periodontology definition.

The two groups were the control group (C group), where surgical peri-implantitis therapy was performed with the use of an access flap and mechanical instrumentation of the contaminated implant surface. In the test group (Laser group), surgical treatment was carried out with the conjunctional use of laser irradiation of the contaminated implant surface.

In order to assess peri-implant osseous defect depth, a radiographic examination was performed at baseline.

The assignment of patients into the two groups of the study was succeeded by a randomization process with the use of computer software (www.randomizer.org). In patients with more than one implant having peri-implantitis, a second randomization procedure with the same procedure determined which implant would be included. The randomization results were placed in opaque envelopes accessible only by the supervisor (I.V.) and given to the treating investigator for each patient, just prior to therapeutic intervention. The present research study was approved by the Ethics Committee of the School of Dentistry. Protocol No. 83/15-06-2020. All participants received written information regarding the aim and the procedures of the study, and afterwards, they were asked to sign their consent.

Sample size calculation was performed on a patient-based analysis in order to detect a clinically significant difference in probing pocket depth (PPD) of 1mm±0.75 mm SD between the two groups (control and laser). Type I error was set at 0.05 level and power at 0.80. The minimum required sample size was calculated to be ten patients per group. In addition, in order to detect a clinically significant difference in PPD of 1mm±1mm SD between the two time periods, within the group, with 0.05 type I error and 0.80 power, the minimum required sample size was estimated to be ten patients per group too.

Treatment Timeline:

After an initial clinical and radiographic examination, patients were screened, and accordingly, suitability for enrollment in the study was confirmed. At the baseline examination, clinical measurements, and peri-implant crevicular fluid (PICF) collection for biomarker sampling were performed. The PICF was retrieved prior to probing and at least 24h after the initial examination to avoid contamination with blood. At the baseline session, after the initial assessment, patients received oral hygiene indications and non-surgical therapy of peri-implant defects in terms of scaling and root planing with titanium curettes and the adjunctive use of chlorhexidine 0.20% irrigation of the peri-implant sulcus. Mechanical debridement using ultrasonics and hand instruments was also performed on the whole dentition prior to surgery. Four-six weeks after the non-surgical treatment the surgery was scheduled. Each patient was followed up for two weeks, three months, and six months post-surgically, and an oral hygiene reinforcement was performed. Clinical measurements and biomarker evaluations were conducted at baseline and six months post-surgically. The following clinical parameters were recorded at baseline and six months after treatment: Full-mouth plaque score (FMPS), percentage of sites positive on bleeding on probing (BoP), probing pocket depth (PPD), gingival recession (REC), and probing attachment levels (PAL).

* BoP: presence (+) or absence (-) of bleeding in percentage (%) 30 s after probe insertion in the peri-implant pocket
* FMPS: Full-Mouth plaque score
* PPD: the distance from the mucosa margin to the bottom of the peri-implant pocket.
* REC: the distance from the prosthetic crown shoulder to the mucosa margin
* PAL: the distance from the prosthetic crown shoulder to the bottom of the sulcus or the peri-implant pocket.

All measurements were recorded at six sites per implant with a 15-mm scale periodontal probe and graded per 1 mm (Hu-friedy® CP-12). The three deepest sites at each implant were included in the statistical analysis for PPD and PAL assessment. All the examinations were performed by the same examiner (I.F.). Intra-examiner reproducibility was calculated during two calibration sessions. Intra-examiner agreement was assessed with an intraclass correlation coefficient (ICC) and showed an agreement of 0.93 (95% CI: 0.89 to 0.96).

Surgical Procedures Local anesthesia was applied, and each patient used a mouthwash solution of 0.20 % chlorhexidine for presurgical mouth disinfection. After an internal bevel incision, full-thickness flaps were raised to access the peri-implant osseous defects.

* Control Group (Group C): removal of granulation tissue and mechanical instrumentation of the implant surface with the use of titanium implant scalers (@Hu-Friedy, IMPLG1/2T) were performed. The instrumentation was followed by thorough cleansing of the implant surface using sterilized gauze soaked in chlorhexidine 0,2% solution.
* Test Group (Group L): In the test group, Nd: YAG laser, 1064nm (Fotona, Light Walker AT, Ljubljana, Slovenia) combined with Er: YAG laser,2940nm (Fotona, Light Walker AT, Ljubljana, Slovenia) was used. Initially, granulation tissue removal was performed by utilizing Er: YAG laser 160mJ, 10Hz, LP, 1.3mm cylindrical tip, handpiece H14-C, W/A:6/4, 30ml per minute. Additionally, decontamination of the implant surface was performed with Er: YAG laser 2940nm, QSP mode, 45mj, 20Hz, non-contact, handpiece H02-C, W/A: 6/4 . Bleeding spots and bone disinfection were created with the application of Εr: YAG laser 160mJ, 15Hz, non-contact, H02-C handpiece, W/A: 6/4 (Fotona, Light Walker AT, Ljubljana, Slovenia). Following that, the Nd: YAG laser 1,5W, 15Hz, MSP, non-contact R21-C3 handpiece, 300μm fiber was applied for deep tissue decontamination and microbial load reduction. Care was taken for the fiber not to aim at the implant surface. Finally, Nd: YAG laser 0,5W, 10Hz, VLP, non-contact R21-C3 handpiece, 300μm fiber (Fotona, Light Walker AT, Ljubljana, Slovenia) in low level was applied after suturing for photobiomodulation. All laser settings were based on the Laser's physical properties and interaction with tissues and implant surfaces. The protocol was planned in cooperation with the laser company considering previous studies using Er: YAG lasers in peri-implantitis . During the laser radiation, both the dental staff and the patients were wearing protective glasses. In both the control and laser group, osteoplasty was performed when needed for better flap adaptation.

The endpoint of debridement for each treatment was determined by macroscopic inspection of the defect site. After suturing, post-surgical instructions, and analgesics (ibuprofen 400 mg three times a day for four days) were administered to the patients. The sutures were removed about 14 days after surgery, and post-surgical instructions were given to all patients. These included a chlorhexidine 0.12 % mouth rinse twice a day for two weeks, for the control group only, and careful tooth brushing with a soft toothbrush so that the sutured area was efficiently cleaned but not traumatized for both groups.

Biomarker's collection and evaluation Peri-implant crevicular fluid (PICF) and samples were collected from one implant site of each individual participating in the study. The specimens were retrieved at least 24 h after the initial clinical examination to avoid contamination with blood from peri-implant sites demonstrating the deepest probing depth. The samples were retrieved using the filter paper technique. In brief, the sampling sites were isolated, air dried, and isolated with cotton rolls supra-gingival biofilm was gently removed, and then a fine, sterile paper strip was inserted into the peri-implant sulcus/pocket until mild resistance was felt and left in place for 30s. Strips that were visually contaminated with blood or saliva were discarded. The obtained sampled fluid volume in the strip was measured by calculating the resorbed PICF volume per 30s, and the paper strips were inserted in micro-centrifuge plastic tubes. The obtained samples were stored at -80°C until being processed for biochemical analysis by enzyme-linked immunosorbent assays (ELISA).

Before the analysis, the samples were diluted with phosphate buffer solution (PBS), centrifuged for 20 min at 4000 g to separate the cells and debris, and then the paper strips were removed. The obtained samples were stored at 20°C until being processed for biochemical analysis. Commercially available ELISA kits were used to measure the concentrations of the bone biomarkers: sRANKL and OPG, from the PICF (Biovendor sRANKL (total) Human ELISA (Osteoprotegerin Ligand, OPG (total) Human Osteoprotegerin, Biovendor - Labolatorni medicina a.s - Czech Republic). The minimal detection limits were: sRANKL (0.4 pmol/l), and OPG (0.03 pmol/l). The ELISA in brief and the monoclonal antibodies specific for these biomarkers were pre-coated into a micro-plate. After washing off unbound substances, an enzyme-linked polyclonal antibody specific to the biomarker was added to each well. The plate was incubated at room temperature for 1 hour and the wells were re-washed. After one hour of incubation, a stop solution was added, and the reaction was arrested. The color developed, being proportional to the amount of biomarker bound in the initial step, allowed measuring its intensity using spectrophotometry (450/620 nm, ELISA processor). A calibration curve was plotted by regression analysis, and the optical density of the sample was used to estimate the concentration of the biomarkers. The concentrations were expressed as biomarker per 30 seconds (pg/30s). During the laboratory analysis, the samples were blind to the lab technician.

ELIGIBILITY:
The inclusion criteria for patients to participate in the study, indicating the existence of peri-implantitis are based on the most recent case definition of peri-implantitis, i.e.:

* Probing depths of ≥6 mm,
* Bone levels ≥3 mm apical of the most coronal portion of the intraosseous part of the implant, and
* the simultaneous presence of bleeding on probing and/or suppuration
* Implants should be loaded for >12 months.

As exclusion criteria were set :

* A severe systematic disease of patients by which a surgical procedure cannot be performed (e.g., bleeding disorders, uncontrolled diabetes mellitus, etc.),
* treatment of peri-implantitis within the previous 12 months,
* antibiotic intake in the last three months before treatment and
* prosthetic loading of implants > 12 months.
* In addition, peri-implantitis lesions indicated for regeneration (3-walled, craters were excluded from the study and were treated accordingly).

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
Probing Pocket Depth | 6 months
  Clinical Periodontal Marker PPD: the distance from the mucosa margin to the bottom of the peri-implant pocket in mm, measured with a periodontal probe

SECONDARY OUTCOMES:
Probing Attachment Levels | 6 months
  Clinical Periodontal Marker: The distance from the implant neck to the bottom of the bottom of the peri-implant pocket measured in mm
Bleeding On Probing | 6 months
  Clinical Periodontal Marker: Bleeding after slight pressure of the mucosal margin with a periodontal probe
Bone loss Biomarkers RANKL/OPG | 6 months
  Rankl and Opg are proteins responsible for bone remodeling. Their ratio is indicative of bone loss or gain. The biomarker is meausured from the peri-implant fluid based on enzyme - immunoabsorbanse test (ELISA)

CONTACTS AND LOCATIONS:
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Makedonia, Greece